CLINICAL TRIAL: NCT06637501
Title: A Multicenter, Open-Label, Phase 2 Study to Investigate the Efficacy and Safety of Sonrotoclax Combined With Zanubrutinib Compared With Zanubrutinib Monotherapy in Adult Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study to Investigate Sonrotoclax Combined With Zanubrutinib Versus Zanubrutinib Alone in Participants With Previously Untreated Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-204; 2024-513970-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Combination Therapy: Sonrotoclax + Zanubrutinib (Experimental): Participants will receive sonrotoclax in combination with zanubrutinib daily for a fixed duration of 15 cycles.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Arm B: Monotherapy: Zanubrutinib (Active Comparator): Participants will receive zanubrutinib monotherapy daily until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
  Arms: Arm A: Combination Therapy: Sonrotoclax + Zanubrutinib
Drug: Zanubrutinib — Administered orally
  Other Names: BRUKINSA; BGB-3111

SUMMARY:
The purpose of this study is to support the registration plan of sonrotoclax plus zanubrutinib treatment in participants with previously untreated CLL. This study is designed to assess the contribution of sonrotoclax to the efficacy outcome of the combination of zanubrutinib and sonrotoclax.

DETAILED DESCRIPTION:
This study will test how effective and safe Sonrotoclax plus Zanubrutinib treatment compared with Zanubrutinib alone in participants with previously untreated chronic lymphocytic leukemia (CLL).

The main goals of the study are to determine how many participants may no longer have evidence of cancer or have some improvement in the signs and symptoms of cancer after treatment and to determine what adverse events, or side effects, patients might experience.

Sonrotoclax is an experimental drug that works by blocking a protein called B-cell lymphoma-2 (Bcl-2). This protein helps certain types of blood tumor cells to survive and grow. When Sonrotoclax blocks Bcl-2 it slows down or stops the growth of tumor cells and helps them die. This can lead to improvements in patients with CLL disease.

Zanubrutinib is a commercialized product that works by blocking a protein called Bruton's tyrosine kinase (BTK) and controlling the activity and survival of malignant B cells. Zanubrutinib has received approval in over 65 countries/regions worldwide for the treatment of adult participants with B cell malignancies, including CLL.

The study will enroll approximately 87 participants who will be randomly assigned by a computer program to receive one of the following treatments: sonrotoclax + zanubrutinib or zanubrutinib.

The study will take place at multiple centers worldwide. The overall time to participate in this study is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated adult patient ≥ 18 years with a confirmed diagnosis of CLL.
2. CLL requiring treatment as per pre-defined criteria.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2.
4. Measurable disease by CT/MRI.
5. Adequate marrow function.
6. Adequate liver function as indicated by aspartate aminotransferase (AST) alanine aminotransferase (ALT) and serum total bilirubin.
7. Adequate renal function.
8. Life expectancy > 6 months.
9. Signed informed consent and able to comply with the study protocol in the investigator's judgment.
10. Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 90 days after the last dose of study drug.

Exclusion Criteria:

1. Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
2. Known central nervous system involvement
3. Received previous systemic treatment for CLL
4. Clinically significant cardiovascular disease
5. Severe or debilitating pulmonary disease
6. History of prior malignancy
7. Active fungal, bacterial, and/or viral infection requiring systemic therapy
8. Positive HIV serology (HIVAb) status or serologic status reflecting active hepatitis B or C infection
9. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring treatment
10. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
11. History of stroke or intracranial hemorrhage ≤ 6 months before the first dose of study treatment
12. Unable to swallow capsules or tablets or diseases significantly affecting GI function
13. Hypersensitivity to zanubrutinib, sonrotoclax, or any of its excipients
14. Use of investigational agents within the last 4 weeks before screening
15. Pregnant and lactating females

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR)/ Complete Response with Incomplete Bone Marrow Recovery (CRi) Rate | Month 16
  Best CR/CRi rate per the Independent Review Committee (IRC) response assessment using the 2018 International Workshop on Chronic Lymphocytic Leukemia guidelines with modification for treatment-related lymphocytosis for participants with CLL

SECONDARY OUTCOMES:
Undetectable Minimal Residual Disease at < 10^-4Sensitivity (uMRD4) Rate | Month 16
  uMRD4 rate measured in both peripheral blood and bone marrow aspirate
CR/CRi Rate per Investigator Response Assessment | Month 16
  CR/CRi Rate (CRR) is defined as the proportion of participants with best overall response of CR or CRi
Overall Response Rate (ORR) per IRC and Investigator Response Assessment | Up to 66 Months
  ORR is defined as the proportion of participants achieving overall response (CR+CRi+partial response [PR]+nodular PR) per the IRC and the investigator response assessment.
Landmark Duration of Response Event-free Rate at 12 Months | 66 months
  The 12-month landmark duration of response event-free rate is defined as the proportion of responders who remain alive and progression-free at 12 months since the first determination of response.
Duration of Response (DOR) per Investigator Response Assessment | Up to 66 Months
  DOR is defined as the time from the first determination of response until first documentation of progression or death, whichever occurs first
Time to Response (TTR) per IRC and Investigator Response Assessment | Up to 66 Months
  TTR is defined as the time from treatment initiation to the first documentation of response
Landmark Progression-free Survival Rate at 24 Months per Investigator Assessment | 24 Months
  The 24-month landmark PFS rate is defined as the proportion of participants who remain alive and progression-free at 24 months since the start of treatment
Progression-free Survival (PFS) per Investigator Response Assessment | Up to 66 Months
  PFS is defined as the time from the start of treatment to the first documentation of disease progression or death, whichever occurs first
Overall Survival (OS) | Up to 66 Months
  OS is defined as the time from treatment initiation to death due to any cause
Number of Participants with Adverse Events (AEs) | From first dose of study drug to 30 days after last dose; up to 66 months for Arm A and Arm B
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 and the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) grading scale for hematologic toxicities in CLL Studies as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (33):
- United States (12):
  - Cleveland Clinic Florida, Weston, Florida
  - Northwest Georgia Oncology Centers Marietta, Marietta, Georgia
  - Illinois Cancer Specialists (Niles) Usor, Niles, Illinois
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Nebraska Cancer Specialists (Satellite Site), Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York Cancer and Blood Specialists, Shirley, New York
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - Texas Oncology Dfw, Dallas, Texas
  - Texas Oncology Tyler, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
- Brazil (4):
  - Centro de Pesquisas Oncologicas Cepon, Florianópolis
  - Hospital de Clinicas de Porto Alegre, Porto AlegreRS
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- China (6):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Italy (4):
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Aou Careggi, Servizio Sanitario Toscana, Florence
  - Universita Degli Studi Di Modena Azienda Ospedaliere Policlinco, Modena
  - Aoor Villa Sofia Cervello, Palermo
- Poland (4):
  - Pratia Onkologia Katowice, Katowice
  - Pratia McM Krakow, Krakow
  - Uniwersytecki Szpital Kliniczny Nr W Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny Hematology, Wroclaw
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Cabuenes, Gijón
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/